CLINICAL TRIAL: NCT01005810
Title: A Controlled Trial of N-Acetylcysteine (NAC) in Cannabis Dependent Adolescents
Brief Title: A Trial of N-Acetylcysteine (an Over-the-Counter Medicine) in Adolescents Who Smoke Marijuana
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kevin Gray, MD, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19152; R01DA026777 (NIH)
Record Dates: First submitted 2009-09-10; First posted 2009-11-02 (Estimated); Results first posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Cannabis Dependence
MeSH Terms: conditions — Marijuana Abuse | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-Acetylcysteine (Active Comparator)
  Interventions: Drug: N-Acetylcysteine; Behavioral: Contingency Management
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo; Behavioral: Contingency Management

INTERVENTIONS:
Drug: N-Acetylcysteine — 1200 mg twice daily for 8 weeks
  Other Names: NAC
  Arms: N-Acetylcysteine
Drug: placebo — 2 capsules twice daily for 8 weeks
  Arms: Placebo
Behavioral: Contingency Management — rewarding biologically verified marijuana abstinence during study visits, with an escalating reward schedule

SUMMARY:
This study is investigating how N-Acetylcysteine (NAC), an over-the-counter medication, will reduce marijuana use when combined with Contingency Management, a behavioral treatment. It is hypothesized that marijuana dependent adolescents who are treated with NAC will use less marijuana during treatment when compared to adolescents who receive a placebo.

DETAILED DESCRIPTION:
This protocol involves investigation of N-Acetylcysteine (NAC) as a pharmacological treatment for cannabis dependence in adolescents. While recent advances have been made in psychosocial treatments for cannabis dependent adolescents, minimal work has been done to investigate the potential adjunctive role for pharmacotherapy in treatment. NAC is an inexpensive, over-the-counter agent with a favorable tolerability profile in adults and children, in common use since FDA approval in 1963. Preclinical and preliminary clinical research in adults suggests a role for NAC in addiction treatment via glutamate modulation.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-21 years
* Regular Marijuana smoker meeting DSM-IV criteria for cannabis dependence and seeking marijuana cessation treatment

Exclusion Criteria:

* Allergy or intolerance to NAC
* Pregnancy or lactation
* Use of carbamazepine or nitroglycerine (or any other drug deemed to be hazardous if taken with NAC) within 14 days of study participation
* Current enrollment in treatment for cannabis dependence
* Current substance dependence, other than cannabis or nicotine
* Significant medical or psychiatric illness that may place the participant at increased risk in the judgement of the study physician

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 116 (Actual)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin M Gray, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- N-Acetylcysteine: N-Acetylcysteine : 1200 mg twice daily for 8 weeks
  Contingency Management : rewarding biologically verified marijuana abstinence during study visits, with an escalating reward schedule
- Placebo: placebo : 2 capsules twice daily for 8 weeks
  Contingency Management : rewarding biologically verified marijuana abstinence during study visits, with an escalating reward schedule
Period: Overall Study
Arm/Group | N-Acetylcysteine | Placebo
Started | 58 | 58
Completed | 37 | 33
Not Completed | 21 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N-Acetylcysteine | Placebo | Total
Number analyzed (Participants) | 58 | 58 | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 9 | 18
  Between 18 and 65 years | 49 | 49 | 98
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.9 (1.5) | 18.8 (1.5) | 18.9 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 13 | 32
  Male | 39 | 45 | 84
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 58 | 58 | 116

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Negative Urine Cannabinoid Tests During Treatment
Description: [Total number of negative urine tests per Group divided by the total number of urine tests per Group]*100
Time Frame: weekly during treatment, for 8 weeks
Measure: Number; unit: percentage of negative urine tests
Arm/Group | N-Acetylcysteine | Placebo
Number analyzed (Participants) | 58 | 58
percentage of negative urine tests | 40.9 | 27.2
Statistical Analysis 1: Comparison: N-Acetylcysteine vs Placebo; Test type: Superiority; p = 0.029, Regression, Logistic; Odds Ratio (OR) = 2.35, 95% CI 2-sided [1.05 to 5.24]

ADVERSE EVENTS:
Arm/Group | N-Acetylcysteine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/58
Other Adverse Events (participants affected / at risk) | 24/58 | 27/58
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-Acetylcysteine (N=58) | Placebo (N=58)
Upper Respiratory Infection (Infections and infestations) | 11 (11) | 8 (8)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Decreased appetite (Gastrointestinal disorders) | 1 (1) | 3 (3)
Drowsiness (Nervous system disorders) | 2 (2) | 2 (2)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Insomnia (Psychiatric disorders) | 5 (5) | 8 (8)
Irritability (Psychiatric disorders) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vivid dreams (Psychiatric disorders) | 6 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes